CLINICAL TRIAL: NCT06713096
Title: Prospective and Randomized Study to Evaluate the Impact of the Recovery Pathway on Postoperative Leght of Stay in Coronary Artery Bypass Surgery
Brief Title: Study to Evaluate the Impact of the Recovery Pathway on Postoperative Leght of Stay in Coronary Artery Bypass Surgery
Acronym: KAMAY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 528421059; 50781921600000068 (Registry Identifier: CAAE)
Record Dates: First submitted 2023-11-22; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Enhanced Recovery After Surgery; Quality Improvement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention)
- Interventional care (Active Comparator)
  Interventions: Behavioral: Tempos Certos protocol

INTERVENTIONS:
Behavioral: Tempos Certos protocol — Improve the enhanced recovery by using the Tempos Certos Protocol by the multiprofissional team , using interventions known by science and recommended by scientists.
  Arms: Interventional care

SUMMARY:
This randomized and prospective trial aims to evaluate the implementation of a rapid recovery protocol for coronary artery bypass grafting (CABG) in a hospital serving patients from the Brazilian Unified Health System (Sistema Único de Saúde - SUS). The study will compare outcomes between two groups: patients receiving care under the rapid recovery protocol and those following the standard institutional care.

Primary Objective:

Compare postoperative hospital stay between the rapid recovery group and the usual care group.

Secondary Objectives:

Assess morbidity and mortality between both groups.

Evaluate patient satisfaction using validated tools.

Analyze incremental costs associated with both approaches.

Assess healthcare teams' learning progression regarding the protocol (Kirkpatrick method).

Evaluate adherence to rapid recovery protocol metrics by healthcare teams.

Measure changes in patient safety culture among healthcare professionals.

Hypothesis:

The null hypothesis assumes no difference in hospital stay between the two groups. The alternative hypothesis suggests that the rapid recovery protocol will reduce hospital stay compared to the standard care. Previous findings from Mejia et al. (2022) indicated a 40% reduction in postoperative hospital stay (from 13 to 7.8 days) for cardiac surgery patients under a rapid recovery protocol at the Heart Institute (InCor HCFMUSP).

This trial will provide critical insights into the applicability of enhanced recovery after surgery (ERAS) principles in cardiac surgery within the context of public healthcare, aiming to improve outcomes and optimize resource use.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Undergoing isolated coronary artery bypass grafting (CABG) with elective or urgent status
* Signed informed consent form (ICF)

Exclusion Criteria:

* Emergency patients
* Severe ventricular dysfunction (ejection fraction <30%)
* Renal impairment (creatinine clearance <30 mL/min)
* Atrial fibrillation or need for oral anticoagulation
* Moderate-to-severe anemia (hematocrit <32%)
* STS risk score >4%
* Patient and/or family disagreement with the protocol
* Failure to sign the informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative hospital stay | From admission to the intensive care unit until hospital discharge (an average of 14 days of leght of hospital stay)
  Count of time between admission to the intensive care unit and hospital discharge (in hours and days).

SECONDARY OUTCOMES:
Number of participants with cardiac reoperation, deep sternal wound infection/mediastinitis, stroke, prolonged ventilation, renal failure, or death within 30 days after surgery (morbimortality) | Hospital stay to 30 days after hospital discharge (an average of 14 days of leght of hospital stay)
  Incidence of key morbidities and mortality, including cardiac reoperation, deep sternal wound infection/mediastinitis, stroke, prolonged ventilation, renal failure, and death.
Patient-reported Patient-reported quality of life (SF-36) | Before surgery and 30 days after hospital discharge (an average of 14 days of leght of hospital stay)
  Quality of life assessed by SF-36 survey before surgery and 30 days after hospital discharge. Scores range from 0 to 100, with higher scores indicating better quality of life.
Patient-reported Anxiety and depression (HADS) | Intervention group: Before surgery, at hospital discharge, and 30 days after hospital discharge. Control group: Before surgery and 30 days after hospital discharge (an average of 14 days of leght of hospital stay)
  Assessment of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS). Scores range from 0 to 21 for both anxiety and depression subscales, with higher scores indicating greater levels of anxiety or depression.
Patient experience (HCAHPS) | Between 3 and 30 days after hospital discharge (an average of 14 days of leght of hospital stay).
  Assessment of patient experience using the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) survey.
Incremental Costs Assessed Using Micro-Costing Analysis | From hospital admission through the postoperative period, including readmissions up to 30 days after discharge.
  Incremental costs assessed through a detailed micro-costing analysis of preoperative, intraoperative, and postoperative phases. Costs will include hospital stay (ward and intensive care unit), multiprofessional care, medications (including blood transfusion), surgical room costs (surgery time and equipment), operational equipment, consumables, imaging exams, and medical supplies. Costs associated with readmissions within 30 days after discharge will also be included.

OTHER OUTCOMES:
Kirkpatrick Evaluation Model | Levels 1 and 2: Before training, after training (5 pilot cases conducted in year 1), and at study conclusion. Level 3: After pilot cases (year 1) and study conclusion. Level 4: At study conclusion.
  Assessment of healthcare professionals' training and behavioral changes using the four levels of the Kirkpatrick Evaluation Model:
  Level 1 (Reaction): Assessed participant satisfaction/motivation via a 5-question Likert scale survey (3-point scale: strongly agree, partially agree, strongly disagree) at three time points: before the project, after training and five pilot cases, and after completing randomized recruitment.
  Level 2 (Learning): Evaluated knowledge improvement through a questionnaire (7 multiple-choice questions and 3 true/false questions) at the same time points as Level 1.
  Level 3 (Behavior): Measured adherence to protocol metrics after five pilot cases and at the conclusion of randomized recruitment. Minimum adherence target: 70%.
  Level 4 (Results): Assessed project outcomes, specifically a 40% reduction in postoperative hospital stay with 70% protocol adherence at the end of randomized recruitment.
Patient Safety Culture (HSPSC) | Before training, after training and experience with five pilot cases (first year of the study), and at the conclusion of randomized recruitment.
  Evaluation of patient safety culture among healthcare professionals using the Hospital Survey on Patient Safety Culture (HSPSC), comprising 42 items across 12 dimensions:
  Teamwork within units Organizational learning/continuous improvement Supervisor/manager expectations/actions promoting safety Hospital management support for patient safety Overall perception of safety Feedback and communication about error Communication openness Frequency of event reporting Teamwork across units Staffing Handoffs and transitions Non-punitive response to errors
  Responses will be collected on a 5-point Likert scale ranging from "strongly disagree" or "never" to "strongly agree" or "always." Scores will be classified into three categories:
  Strengthened areas (≥75% positive responses) Potential improvement areas (<75% and >50% positive responses) Fragile areas (≤50% positive responses)

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle B Borgomoni, bsc, PhD student, Principal Investigator — Instituto do coração
Locations (1):
- Hc Da Fmusp Instituto Do Coracao Incor Sao Paulo, São Paulo, São Paulo, Brazil